CLINICAL TRIAL: NCT01726452
Title: Neo-AEGIS (NEOadjuvant Trial in Adenocarcinoma of the oEsophagus and oesophagoGastric Junction International Study): Randomised Clinical Trial of Neoadjuvant and Adjuvant Chemotherapy (Modified MAGIC or FLOT Regimen) vs. Neoadjuvant Chemoradiation (CROSS Protocol) in Adenocarcinoma of the Oesophagus and Oesophago-gastric Junction
Brief Title: NEOadjuvant Trial in Adenocarcinoma of the oEsophagus and oesophagoGastric Junction International Study (Neo-AEGIS)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cancer Trials Ireland (Network)
Collaborators: Southampton Clinical Trials Unit (Unknown); Rigshospitalet, Denmark (Other); Centre Hospitalier Régional, Universitaire de Lille (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTRIAL-IE (ICORG) 10-14
Record Dates: First submitted 2012-11-06; First posted 2012-11-15 (Estimated); Last update posted 2022-09-30 (Actual); Status verified 2022-09

CONDITIONS: Adenocarcinoma of the Oesophagus; Adenocarcinoma of the Oesophago-gastric Junction; Oesophageal Tumours; Junctional Tumours; Oesophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Epirubicin; Cisplatin; Oxaliplatin; Capecitabine; Paclitaxel; Carboplatin; Docetaxel; Leucovorin; Fluorouracil

ARMS (2):
- A (Modified MAGIC) OR Arm A: FLOT (Experimental): Modified MAGIC: The modified MAGIC regimen encompasses 3 cycles of chemotherapy pre-surgery and 3 cycles post-surgery. The regimen is a combination of epirubicin, cisplatin or oxaliplatin and a choice of 5-fluorouracil or capecitabine. Each cycle lasts 21 days.
  FLOT: The FLOT regimen encompasses 8 cycles of chemotherapy in total , 4 cycles of chemotherapy pre-surgery and a further 4 cycles of chemotherapy post-surgery. Each cycle of chemotherapy lasts 14 days/2 weeks.
  Interventions: Drug: Epirubicin; Drug: Cisplatin / Oxaliplatin; Drug: 5 Flourouracil/ Capecitabine; Drug: Docetaxel; Drug: Oxaliplatin; Drug: Leucovorin; Drug: 5-Fluorouracil
- B (CROSS) (Experimental): Arm B consists of the multimodal CROSS arm, which includes a combination of chemotherapy and radiotherapy prior to surgery. The patient will receive four and a half (4.5) weeks of radiation therapy (41.4 Gy/23 fractions), and 5 weekly cycles of chemotherapy. The chemotherapy and radiotherapy will run concurrently over a 4 and a half-week period. Chemotherapy is given by intravenous infusion on days 1, 8, 15, 22 and 29. The radiation will generally commence on the 1st day of treatment and will run for 4 and a half weeks as follows: days 1-5, days 8-12, days 15-19, days 22-26 and days 29-31 inclusive.
  Interventions: Radiation: (41.4 Gy/23 fractions); Drug: Paclitaxel; Drug: Carboplatin

INTERVENTIONS:
Drug: Epirubicin — 50mg/m2 on Day 1 of each cycle only (i.e. every 21 days)
  Arms: A (Modified MAGIC) OR Arm A: FLOT
Drug: Cisplatin / Oxaliplatin — Cisplatin, 60mg/m2 on day 1 of each cycle only (i.e. every 21 days). OR Oxaliplatin,130 mg/m2 on Day 1 of each cycle (i.e. every 21 days) The choice between administering Cisplatin or Oxaliplatin is at the discretion of the investigator.
  Arms: A (Modified MAGIC) OR Arm A: FLOT
Drug: 5 Flourouracil/ Capecitabine — 5-Flourouracil 200 mg/m2/day every day for 21 days OR Capecitabine 625 mg/m2 twice daily orally). The choice between administering 5 Flourouracil or Capecitabine is at the discretion of the investigator.
  Arms: A (Modified MAGIC) OR Arm A: FLOT
Radiation: (41.4 Gy/23 fractions) — Patient will receive 4.5 weeks of radiation therapy (41.4 Gy/23 fractions).
  Arms: B (CROSS)
Drug: Paclitaxel — 50mg/ m2 Paclitaxel dose administered on Days 1, 8, 15,22 and 29. Dexamethasone, Chlorphenamine and Ranitidine dose given per local standard practice. NACL infusion per local standard practice. Ondansetron dose given per local standard practice on Days 1, 8, 15, 22 and 29.
  Arms: B (CROSS)
Drug: Carboplatin — Dose determined as per calculation, infused on Days 1, 8, 15, 22 and 29
  Arms: B (CROSS)
Drug: Docetaxel — Docetaxel, 50 mg/m², day 1 of each cycle (i.e. every 14 days)
  Arms: A (Modified MAGIC) OR Arm A: FLOT
Drug: Oxaliplatin — 85 mg/m², day 1 of each cycle (i.e. every 14 days)
  Arms: A (Modified MAGIC) OR Arm A: FLOT
Drug: Leucovorin — 200 mg/m², day 1 of each cycle (i.e. every 14 days).
  Arms: A (Modified MAGIC) OR Arm A: FLOT
Drug: 5-Fluorouracil — 2600 mg/m² Day 1 of each cycle (i.e. every 14 days) Dexamethasone or equivalent, 8mg, twice daily, Day before, day of and day after OR administered as per standard practice
  Arms: A (Modified MAGIC) OR Arm A: FLOT

SUMMARY:
This is a multicentre phase III open-labelled, randomised controlled trial. Eligible patients will be randomised in a 1:1 fashion between neoadjuvant and adjuvant chemotherapy (Investigator's choice modified MAGIC (ECF/ECX or EOF/EOX) or FLOT regimen) and surgery or Arm B (CROSS protocol: chemotherapy with radiation therapy and surgery as per multimodal protocol).

Primary Objective:

To evaluate one, two and three year survival of patients treated with resection plus neoadjuvant and adjuvant chemotherapy versus resection plus neoadjuvant chemo radiotherapy.

Secondary Objective(s):

To evaluate the effect of both neoadjuvant regimens on clinical and pathological response rate (in particular relief of dysphagia, improvement in health related quality of life (HRQL), endoscopic regression, and CT-PET evidence of tumour response), tumour regression grade, node-positivity, post-operative pathology, disease-free survival, time to treatment failure, toxicity, post-operative complications and Health Related Quality of Life (HRQL).

Exploratory Objective(s):

Translational Research: The collection of blood and tissue samples for storage in the bio bank for future research.

DETAILED DESCRIPTION:
Indication:

Patients with cT2-3 N0-1 M0 adenocarcinoma of the oesophagus or junction, based on clinical, CT-PET, and EUS staging, will be randomised to the modified MAGIC (ECF/ECX or EOF/EOX) or FLOT regimen and chemotherapy regimen versus the CROSS neoadjuvant chemo radiation protocol prior to surgery. Patients will be randomised to either Arm A (modified MAGIC or FLOT chemotherapy only and surgery) or Arm B (CROSS protocol: chemotherapy with radiation therapy and surgery as per multimodal protocol).

Eligible patients will be randomised in a 1:1 fashion between the modified MAGIC or FLOT regimen or the CROSS protocol.

Exploratory Study- Translational Research :

The collection of blood and tissue samples for storage in the bio bank for future research.

Patients enrolled in this trial at the St James's' Hospital site, will be invited to consent to having some of their tissue and blood taken for use in future research studies. Following consent from the patient, tissue biopsy of tumour and/or normal oesophageal tissue will be obtained for research at the same time as that biopsied for histological diagnosis. In addition, tumour and/or normal tissue will also be obtained following surgical resection. Patient blood samples will also be obtained, both before and during treatment. The identification of both tumour and circulating biomarkers will increase knowledge of the molecular mechanism(s) underlying treatment response in oesophageal cancer and may facilitate the identification of biomarkers predicting patient response to treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically verified adenocarcinoma of the oesophagus or oesophago-gastric junction based on endoscopy (OGD)
2. CT-18FDG-PET performed in all patients for disease staging.
3. EUS in all patients unless luminal obstruction precludes sensitivity of the test.
4. Staging laparoscopy performed at the investigator's discretion for locally advanced AEG II and AEG III tumours .
5. Pre-treatment stage cT2-3, N0-3, M0.
6. Maximum tumour length should be no more than 8cm (equal to 8 cm is acceptable)
7. Male/female patients aged ≥18 years
8. ECOG Performance Status 0, 1 or 2 (Appendix F).
9. ASA I-II (Appendix F).
10. Adequate cardiac function. For all patients, an ejection fraction of > 50% is required. If patients have a known cardiac history (e.g. known ischemic disease, cardiomyopathy) an ejection fraction > 50% and cardiac clearance by a consultant cardiologist for major surgery and cancer therapies is required.
11. Adequate respiratory function. Patients should have pulmonary function tests completed with a minimum FEV1 ≥ 1.5L. CPEX acceptable
12. Adequate bone marrow function: absolute neutrophil count (ANC) >1.5x109/l; white blood cell count >3x109/l; platelets >100x109/l; haemoglobin (Hb) >9g/dl (can be post-transfusion).
13. Adequate renal function: glomerular filtration rate >60ml/minute calculated using the Cockcroft-Gault Formula (Appendix O).
14. Adequate liver function: serum bilirubin <1.5x ULN; AST <2.5x ULN and ALP <3x ULN (ULN as per institutional standard).
15. Written informed consent must be obtained from the patient before any study-trial specific procedures are performed.
16. Women of child-bearing potential and male subjects must agree to use an effective barrier method of contraception for up to 6 months following discontinuation of therapy. Effective contraception is defined as any medically recommended (or combination of methods) as per standard of care.
17. Women of childbearing potential must have pregnancy excluded by urine or serum beta-HCG testing within 7 days prior to treatment.

Exclusion Criteria:

1. Tumours of squamous histology.
2. Patients with advanced inoperable or metastatic oesophageal, junctional or gastric adenocarcinoma.
3. Disease length (total length of tumour plus node) greater than 10cm (up to 10 cm will be allowed) -as measured by any modality or, if appropriate, combination of modalities-, unless in the opinion of the investigator in discussion with national RT lead, it is felt that OAR constraints are likely to be achievable.
4. Any prior chemotherapy for gastrointestinal cancer.
5. Prior abdominal or thoracic, chest wall or breast radiotherapy.
6. Patients who are unfit for surgery or cancer treatments based on cardiac disease.
7. Patients with acute systemic infections.
8. Patients who are receiving treatment with sorivudine or its chemical related analogues, such as brivudine which is contraindicated with capecitabine and 5-fluorouracil administration.
9. Clinical COPD with significant obstructive airways disease classified by FEV1 < 1.5 L or PaO2 less than 9kPa on room air
10. Known peripheral neuropathy >Grade 1 (absence of deep tendon reflexes as the sole neurological abnormality does not render the patient ineligible).
11. Known positive tests for human immunodeficiency virus (HIV) infection, acute or chronic active hepatitis B infection.
12. Any other malignancies within the last 5 years (other than curatively treated basal cell carcinoma of the skin and/or in situ carcinoma of the cervix)
13. Participation in other clinical trials of investigational or marketed agents for the treatment of oesophageal cancer or other diseases within 30 days from registration. UK sites please refer to Group Specific Appendix
14. Women who are pregnant or breastfeeding.
15. Psychiatric illness/social situations that would limit compliance with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 377 (Actual)
Dates: Start 2013-01-24 (Actual); Primary Completion 2022-08-04 (Actual); Study Completion 2022-08-04 (Actual)

PRIMARY OUTCOMES:
Overall survival | At end of trial- up to 3 years in follow up
  Overall survival will be calculated from the date of randomisation and an event registered on the date of death from any cause. Patients lost to follow up, or those with no death recorded on the day the database is frozen, will be censored on the date of last follow up.

CONTACTS AND LOCATIONS:
Overall Officials: John V. Reynolds, Professor, Principal Investigator — Trinity Centre, St. James's Hospital, Dublin 8, Ireland
Locations (29):
- Rigshospitalet, Blegdamsvej 9, Denmark
- Centre Hospitalier Régional, Universitaire de Lille 2 Avenue Oscar Lambret, 59000, Lille, France
- Ireland (5):
  - Cork University Hospital, Cork
  - Beaumont Hospital, Dublin
  - SLRON- St Luke's Radiation Oncology Network, Dublin
  - St. James's Hospital, Dublin
  - University Hospital Galway, Galway
- Karolinska Institutet and Karolinska University Hospital, Stockholm, Sweden
- United Kingdom (21):
  - The Royal Bournemouth Hospital, The Royal Bournemouth and Christchurch Hospitals NHS Foundation, Bournemouth
  - Cambridge University Hospitals NHS Foundation Trust, Addenbrooke's Hospital, Box 279(s4), Cambridge Biomedical Camp, Cambridge
  - Velindre Cancer Centre, Velindre NHS Trust, Velindre Road, Whitchurch, Cardiff
  - University Hospitals Coventry & Warwickshire, Clifford Bridge Road, Walsgrave, Coventry
  - Hull and East Yorkshire Hospitals NHS Trust, Castle Hill Hospital,, Cottingham, East Riding Of Yorkshire
  - Portsmouth Hospitals NHS Trust, Southwick Hill Road, Cosham, Hampshire
  - Mount Vernon Cancer Centre, E & N Hertfordshire NHS Trust, Rickmansworth Road, Northwood, Middlesex
  - Nottingham City Hospital, Nottingham University Hospitals NHS Trust, Hucknall Road, Nottingham
  - Oxford University Hospital NHS Trust Churchill Hospital, Headington, Oxfordshire
  - University Hospital Southampton NHS Foundation Trust, Southampton General Hospital, Division A Cancer Care, Mp307, T, Southampton
  - Royal Surrey County Hospital, Guildford, Surrey
  - Worcestershire Royal Hospital, Worcestershire Oncology Centre, Charles Hastings Way, Worcester
  - Belfast Health and Social Care Trust, Northern Ireland Cancer Centre, Belfast CityHospital, Belfast
  - The Clatterbridge Cancer Centre NHS Foundation Trust, Birkenhead, Wirral
  - University Hospitals Bristol NHS Foundation Trust, Bristol
  - University Hospital Plymouth NHS Trust, Derriford Hospital, Derriford Road, Crownhill, Plymouth
  - NHS Lothian, Edinburgh Cancer Centre,, Edinburgh
  - Beatson West of Scotland Cancer Centre, Glasgow, 1056 Great Western Road
  - Imperial College Healthcare NHS Trust St Mary's Hospital, London
  - The Newcastle upon Tyne Hospital NHS Foundation TrustFreeman Hospital, Freeman Road, High Heaton, Newcastle upon Tyne
  - Royal Preston Hospital, Sharoe Garoo Lane, Fulwood, Preston

REFERENCES:
- [Derived] Reynolds JV, Preston SR, O'Neill B, Lowery MA, Baeksgaard L, Crosby T, Cunningham M, Cuffe S, Griffiths GO, Parker I, Risumlund SL, Roy R, Falk S, Hanna GB, Bartlett FR, Alvarez-Iglesias A, Achiam MP, Nilsson M, Piessen G, Ravi N, O'Toole D, Johnston C, McDermott RS, Turkington RC, Wahed S, Sothi S, Ford H, Wadley MS, Power D; Neo-AEGIS Investigators and Trial Group. Trimodality therapy versus perioperative chemotherapy in the management of locally advanced adenocarcinoma of the oesophagus and oesophagogastric junction (Neo-AEGIS): an open-label, randomised, phase 3 trial. Lancet Gastroenterol Hepatol. 2023 Nov;8(11):1015-1027. doi: 10.1016/S2468-1253(23)00243-1. Epub 2023 Sep 18. PMID 37734399
- [Derived] Reynolds JV, Preston SR, O'Neill B, Baeksgaard L, Griffin SM, Mariette C, Cuffe S, Cunningham M, Crosby T, Parker I, Hofland K, Hanna G, Svendsen LB, Donohoe CL, Muldoon C, O'Toole D, Johnson C, Ravi N, Jones G, Corkhill AK, Illsley M, Mellor J, Lee K, Dib M, Marchesin V, Cunnane M, Scott K, Lawner P, Warren S, O'Reilly S, O'Dowd G, Leonard G, Hennessy B, Dermott RM. ICORG 10-14: NEOadjuvant trial in Adenocarcinoma of the oEsophagus and oesophagoGastric junction International Study (Neo-AEGIS). BMC Cancer. 2017 Jun 3;17(1):401. doi: 10.1186/s12885-017-3386-2. PMID 28578652